CLINICAL TRIAL: NCT04376047
Title: Effect of Reverse Trendelenburg Position Versus Semi-recumbent Position on Ventilation and Oxygenation Parameters in Obese Critically Ill Patients: Randomized Controlled Trial
Brief Title: Reverse Trendelenburg Position Versus Semi-recumbent Position in Obese Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1212020
Record Dates: First submitted 2020-04-18; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Ventilation and Oxygenation; Obese; Positioning; Critically Ill
Keywords: Reverse Trendelenburg position; semi-recumbent position; ventilation; oxygenation; obese patients
MeSH Terms: conditions — Respiratory Aspiration; Obesity; Critical Illness

STUDY DESIGN:
Intervention Model Description: two-group pre-test and repeated post-test study
Who Masked: Care Provider
Masking Description: Computer generated randomization (www.randomizer.org) was used to randomly assign patients to one of both groups. Information of allocation was available to the principal researcher only. Patients were assigned a sequential number that was placed in an opaque, sealed envelope by the researcher. When the patients were scheduled to be positioning, the envelope was opened by the researcher who then performed the positioning. The nurses could not be blinded to the allocation because of the nature of the intervention. However, the outcome assessment of the patients was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse Trendelenburg position group (Experimental): Obese critically ill patients who are positioned in reverse Trendelenburg position
  Interventions: Other: Reverse Trendelenburg position
- Semi-recumbent position group (Active Comparator): Obese critically ill patients who are positioned in semi-recumbent position which is the routine ICU position
  Interventions: Other: Semi-recumbent position

INTERVENTIONS:
Other: Reverse Trendelenburg position — The Reverse Trendelenburg position is a position in which patients' hip and knee are not flexed but the head and chest are elevated at 30° than the abdomen and legs.
  Arms: Reverse Trendelenburg position group
Other: Semi-recumbent position — The semi-recumbent position is an upright positioning of the head and torso at an angle of 45° while legs are lying on the bed.
  Arms: Semi-recumbent position group

SUMMARY:
The aim of this study is to assess the effect of reverse Trendelenburg position versus semi-recumbent position on ventilation and oxygenation parameters of obese critically ill patients

DETAILED DESCRIPTION:
Obese critically ill patients' position significantly impacts on their ventilation and oxygenation status. It is also associated with mechanical ventilation success or failure and may be a main determinant of the obese patients' outcome. Reverse Trendelenburg position is recommended for obese patients but in critical illness with mechanical ventilation little is known about its effect on respiratory therapeutic targets. This trial was conducted in four general intensive care unit of Alexandria Main University hospital in Alexandria, Egypt. One hundred and ten adult mechanically ventilated patients with body mass index ≥ 30 were randomly assigned by a computer program to either reverse Trendelenburg position group (n=55) which is the intervention group or semi-recumbent position group (n=55) which is the routine unit position. Patients were positioned in the study positions 4 times per day. Patients were maintained in the study positions for 2 hours each time. Baseline ventilation and oxygenation parameters were assessed immediately before positioning then it was reassessed every 10 minutes after positioning for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 30
* Mechanically ventilated

Exclusion Criteria:

* Trauma
* Shock
* Acute respiratory distress syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Respiratory dynamic compliance | 30 minute form positioning time
  Respiratory dynamic compliance (Cdyn) in ml/cm H2O is the change in lung volume per unit change in pressure in the presence of flow. It is calculated through the equation of tidal volume/ (peak inspiratory pressure - positive end expiatory pressure). All the previous equation variables are assessed from the patient's mechanical ventilator data.
Respiratory minute volume | 30 minute form positioning time
  Respiratory minute volume (VE) in mL/min is the total volume of air that is expired over one minute. It is calculated directly by the mechanical ventilator and presented on patient's mechanical ventilator data.
Partial pressure carbon dioxide | 30 minute form positioning time
  Partial pressure carbon dioxide (PaCO2) in mm Hg is assessed from arterial blood gases sample.
Partial pressure oxygen | 30 minute form positioning time
  Partial pressure oxygen (PaO2) in mm Hg is assessed from arterial blood gases sample.
Hypoxemic index | 30 minute form positioning time
  Hypoxemic index is the ratio of partial pressure oxygen to fraction inspiratory oxygen (PaO2/FiO2).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Researchers are waiting to get approval from research committee to make individual participant data (IPD) available to other researchers